CLINICAL TRIAL: NCT00014859
Title: Epidemiology of Surfactant Protein-B Deficiency
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, F. Sessions Cole, MD, Professor of Pediatrics, Washington University School of Medicine
Other Study IDs: 967; NCT00200915 (obsolete NCT alias)
Record Dates: First submitted 2001-04-11; First posted 2001-04-12 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Lung Diseases; Respiratory Distress Syndrome, Newborn; Pulmonary Surfactant; Lung Diseases, Interstitial
Keywords: Pulmonary surfactant; Surfactant protein B; Surfactant protein C; ABCA3; NKX2-1; Alveolar type 2 cell
MeSH Terms: conditions — Lung Diseases; Respiratory Distress Syndrome, Newborn; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — DNA and tracheal aspirate samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Population-based cohort: Descriptive cohort of population-based DNA samples from the newborn screening program in Missouri with vital statistics based, linked phenotype data
- Trio sequencing cohort: Affected infant/child (term or near term infant with progressive respiratory distress or other rare pulmonary phenotype or older child with interstitial lung disease or other rare pulmonary phenotype) and parents

SUMMARY:
The purpose of this study is to test the hypothesis that excess, rare, functionally disruptive single nucleotide polymorphisms (SNPs) characterize genes (e.g., the surfactant protein-B gene)(SFTPB) and gene networks (e.g., the pulmonary surfactant metabolic network or other gene networks that regulate alveolar type 2 cell function) associated with increased risk of neonatal respiratory distress syndrome (RDS).

DETAILED DESCRIPTION:
BACKGROUND:

Respiratory distress syndrome is the most frequent respiratory cause of death and morbidity in infants less than 1 year of age in the United States. Of approximately 28,500 infant deaths in 2006, 5,421 (19.7%) were diagnosed with respiratory distress as either the primary (1,011 - 3.7%) or secondary (4,410 - 16%) cause of death. Despite improvement in infant mortality rates over the last 20 years, survivors of respiratory distress syndrome with chronic respiratory disease consume twenty times more annualized dollars than unaffected children and 5.9% of all dollars spent on children from 0-18 years of age. More recent estimates including data from California and New York, the Institute of Medicine, and the 2001 Nationwide Inpatient Sample from the Healthcare Cost and Utilization Project suggest that the average cost of hospitalization for each of the 49,900 infants with a diagnosis of respiratory distress syndrome was $56,800 vs. $10,700 for a premature infant without respiratory distress syndrome. The recent increase in late preterm births has contributed to both the frequency of respiratory distress syndrome and its economic impact. These medical costs do not include the economic consequences of infant respiratory morbidity for families, e.g., absence from work, and early intervention costs to optimize outcome. In addition, despite 2-3 fold greater risk of infant mortality for African American infants than European American infants from all other causes, European American infants have greater risk of death from respiratory distress than African American infants, and this increased risk is not attributable to differences in surfactant phospholipid composition, birth weight, gestational age, or confounding socioeconomic factors. Understanding the genetic mechanisms that cause respiratory distress syndrome is critical for improving outcomes of children in the United States, reducing costs of their health care, and reducing racial disparity in infant mortality. Since the original description of deficiency of the pulmonary surfactant in premature newborn infants by Avery and Mead in 1959, respiratory distress syndrome has most commonly been attributed to developmental immaturity of pulmonary surfactant production. Despite improvement in neonatal survival associated with availability of surfactant replacement therapy for premature infants, gender and race based disparities in disease frequency, morbidity and mortality have persisted, an observation that suggests that genetic factors play an important role in disease pathogenesis. In addition, twin studies indicate high heritability (h2) of neonatal respiratory distress syndrome (0.2 and 0.8). Recent clinical reports of monogenic causes of neonatal respiratory distress syndrome, statistical association of candidate gene variants with increased disease risk, and studies of targeted gene ablation in murine lineages have also strongly suggested that genetic mechanisms contribute to risk of respiratory distress syndrome in newborn infants. When we examined genetic variants in large population-based and case-control cohorts, we found that the population-based frequencies of individual, disruptive mutations in 3 candidate genes (SFTPB, SFTPC, and ABCA3) (<2%) account for <0.1% of the population attributable risk in term or near term infants, and that individual, rare, disruptive mutations are not associated with disease in case-control cohorts. In addition, when we attempted to establish an association between an intermediate biochemical phenotype (surfactant protein-B peptide mobility on western blot) and SFTPB variants (assessed by complete resequencing) in term and near term infants with and without respiratory distress, we failed to identify a SFTPB variant or combination of variants associated with respiratory distress and altered surfactant protein-B structure. Finally, we have recently found that tagSNPs in genes from gene networks expressed in lung but not part of the pulmonary surfactant network (ion channel, lung remodeling, and unfolded protein response genes) confer race-specific risk of neonatal respiratory distress syndrome. These studies suggest that variation in SFTPB, SFTPC, and ABCA3 is under significant purifying selection pressure and that the genetic contribution to neonatal respiratory distress syndrome is based on contributions of rare, independent risk alleles in multiple genes and gene networks.

DESIGN NARRATIVE:

Rare mutations in the surfactant protein-B gene (SFTPB) and other genes in the pulmonary surfactant metabolic network cause lethal neonatal respiratory distress syndrome in human newborn infants by disrupting metabolism and function of the pulmonary surfactant. Mutation frequencies (<1-2%) in SFTPB and 2 other candidate genes in the pulmonary surfactant network (SFTPC and ABCA3) do not account for heritability of neonatal respiratory distress syndrome (h2~0.2-0.8) suggested by twin studies. To develop a comprehensive catalogue of genes and gene networks that account for the heritability of this complex disease, we propose to test the hypothesis that excess, rare, functionally disruptive single nucleotide polymorphisms (SNPs) characterize genes and gene networks associated with increased risk of neonatal respiratory distress syndrome. Specifically, using trio whole exome or whole genome sequencing of affected infant (progressive, severe respiratory distress in term or near term infants or children with unexplained interstitial lung disease or other rare lung phenotypes)/parent trios, we will identify de novo or recessively inherited pathogenic variants including single nucleotide variants, small insertions/deletions, and copy number or structural variants (>100 kb). To predict pathogenicity, we will use a suite of computational prediction algorithms (e.g., ANNOVAR, CADD). To confirm variants in genes and gene pathways not previously associated with human infant/child rare respiratory phenotypes, we will use GeneMatcher to identify other affected infants with pathogenic variants at the same gene locus or in the same gene pathway or functional testing of identified variants in a variety of cell-based jor model organism models. Using next-generation sequencing technology and state of the art statistical methods to elucidate the genetic complexity of neonatal respiratory distress syndrome and rare infant lung phenotypes will permit the development of personalized diagnostic tools and preventive therapeutic strategies for high risk infants and young children.

ELIGIBILITY:
Inclusion Criteria:

* Normal pulmonary function or a diagnosis of RDS

Exclusion Criteria:

* None

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cohort I is a population-based cohort from Missouri. Cohort II is a cohort of family trios (affected infant/child and parents) which may also include other unaffected or affected siblings from the Neonatal Intensive Care Unit at St. Louis Children's Hospital and from patients referred from other centers.
Sampling Method: Non-Probability Sample
Enrollment: 5176 (Actual)
Dates: Start 2001-06-01 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Statistical association of rare, functionally disruptive genomic variant with RDS | 4 weeks
  Using trio whole exome or whole genome sequencing, next generation sequencing, and in silico prediction of function, discover statistical associations between gene loci with excess, rare, functionally disruptive variants and risk of neonatal respiratory distress syndrome.

SECONDARY OUTCOMES:
Statistical associations between risk of neonatal respiratory distress syndrome and excess, rare functional variants in gene pathways | 4 weeks
  Using trio whole exome or whole genome sequencing, next generation sequencing, in silico prediction of functional variants, and Metacore for pathway construction, identify statistical associations between risk of neonatal respiratory distress syndrome and pathways with excess, rare functional variants

CONTACTS AND LOCATIONS:
Overall Officials: F. Sessions Cole, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
All new variants will be deposited in public databases immediately after publication.

REFERENCES:
- [Background] Merchak A, Janssen DJ, Bohlin K, Patterson BW, Zimmermann LJ, Carnielli VP, Hamvas A. Endogenous pulmonary surfactant metabolism is not affected by mode of ventilation in premature infants with respiratory distress syndrome. J Pediatr. 2002 Jun;140(6):693-8. doi: 10.1067/mpd.2002.124320. PMID 12072872
- [Background] Nogee LM. Genetic mechanisms of surfactant deficiency. Biol Neonate. 2004;85(4):314-8. doi: 10.1159/000078171. Epub 2004 Jun 8. PMID 15218289
- [Background] Cameron HS, Somaschini M, Carrera P, Hamvas A, Whitsett JA, Wert SE, Deutsch G, Nogee LM. A common mutation in the surfactant protein C gene associated with lung disease. J Pediatr. 2005 Mar;146(3):370-5. doi: 10.1016/j.jpeds.2004.10.028. PMID 15756222
- [Background] Kingsmore SF, Cole FS. The Role of Genome Sequencing in Neonatal Intensive Care Units. Annu Rev Genomics Hum Genet. 2022 Aug 31;23:427-448. doi: 10.1146/annurev-genom-120921-103442. Epub 2022 Jun 8. PMID 35676073
- [Background] Wambach JA, Nogee LM, Cole FS. First Steps toward Personalized Therapies for ABCA3 Deficiency. Am J Respir Cell Mol Biol. 2022 Apr;66(4):349-350. doi: 10.1165/rcmb.2021-0405ED. No abstract available. PMID 35077664
- [Result] Nogee LM. Abnormal expression of surfactant protein C and lung disease. Am J Respir Cell Mol Biol. 2002 Jun;26(6):641-4. doi: 10.1165/ajrcmb.26.6.f241. No abstract available. PMID 12034561
- [Result] Cole FS. Surfactant protein B: unambiguously necessary for adult pulmonary function. Am J Physiol Lung Cell Mol Physiol. 2003 Sep;285(3):L540-2. doi: 10.1152/ajplung.00111.2003. No abstract available. PMID 12902317
- [Result] Hamvas A, Madden KK, Nogee LM, Trusgnich MA, Wegner DJ, Heins HB, Cole FS. Informed consent for genetic research. Arch Pediatr Adolesc Med. 2004 Jun;158(6):551-5. doi: 10.1001/archpedi.158.6.551. PMID 15184218
- [Result] Hamvas A, Nogee LM, White FV, Schuler P, Hackett BP, Huddleston CB, Mendeloff EN, Hsu FF, Wert SE, Gonzales LW, Beers MF, Ballard PL. Progressive lung disease and surfactant dysfunction with a deletion in surfactant protein C gene. Am J Respir Cell Mol Biol. 2004 Jun;30(6):771-6. doi: 10.1165/rcmb.2003-0323OC. Epub 2003 Dec 4. PMID 14656744
- [Result] Hamvas A, Wegner DJ, Trusgnich MA, Madden K, Heins H, Liu Y, Rice T, An P, Watkins-Torry J, Cole FS. Genetic variant characterization in intron 4 of the surfactant protein B gene. Hum Mutat. 2005 Nov;26(5):494-5. doi: 10.1002/humu.9378. PMID 16211553
- [Result] Palomar LM, Nogee LM, Sweet SC, Huddleston CB, Cole FS, Hamvas A. Long-term outcomes after infant lung transplantation for surfactant protein B deficiency related to other causes of respiratory failure. J Pediatr. 2006 Oct;149(4):548-53. doi: 10.1016/j.jpeds.2006.06.004. PMID 17011330
- [Result] Cole FS, Nogee LM, Hamvas A. Defects in surfactant synthesis: clinical implications. Pediatr Clin North Am. 2006 Oct;53(5):911-27, ix. doi: 10.1016/j.pcl.2006.08.006. PMID 17027617
- [Result] Wilson RK, Ley TJ, Cole FS, Milbrandt JD, Clifton S, Fulton L, Fewell G, Minx P, Sun H, McLellan M, Pohl C, Mardis ER. Mutational profiling in the human genome. Cold Spring Harb Symp Quant Biol. 2003;68:23-9. doi: 10.1101/sqb.2003.68.23. No abstract available. PMID 15338599
- [Result] Wegner DJ, Hertzberg T, Heins HB, Elmberger G, MacCoss MJ, Carlson CS, Nogee LM, Cole FS, Hamvas A. A major deletion in the surfactant protein-B gene causing lethal respiratory distress. Acta Paediatr. 2007 Apr;96(4):516-20. doi: 10.1111/j.1651-2227.2006.00188.x. PMID 17391469
- [Result] Hamvas A, Wegner DJ, Carlson CS, Bergmann KR, Trusgnich MA, Fulton L, Kasai Y, An P, Mardis ER, Wilson RK, Cole FS. Comprehensive genetic variant discovery in the surfactant protein B gene. Pediatr Res. 2007 Aug;62(2):170-5. doi: 10.1203/PDR.0b013e3180a03232. PMID 17597650
- [Result] Saugstad OD, Hansen TW, Ronnestad A, Nakstad B, Tollofsrud PA, Reinholt F, Hamvas A, Coles FS, Dean M, Wert SE, Whitsett JA, Nogee LM. Novel mutations in the gene encoding ATP binding cassette protein member A3 (ABCA3) resulting in fatal neonatal lung disease. Acta Paediatr. 2007 Feb;96(2):185-90. doi: 10.1111/j.1651-2227.2007.00016.x. PMID 17429902
- [Result] Garmany TH, Wambach JA, Heins HB, Watkins-Torry JM, Wegner DJ, Bennet K, An P, Land G, Saugstad OD, Henderson H, Nogee LM, Cole FS, Hamvas A. Population and disease-based prevalence of the common mutations associated with surfactant deficiency. Pediatr Res. 2008 Jun;63(6):645-9. doi: 10.1203/PDR.0b013e31816fdbeb. PMID 18317237
- [Result] McBee AD, Wegner DJ, Carlson CS, Wambach JA, Yang P, Heins HB, Saugstad OD, Trusgnich MA, Watkins-Torry J, Nogee LM, Henderson H, Cole FS, Hamvas A. Recombination as a mechanism for sporadic mutation in the surfactant protein-C gene. Pediatr Pulmonol. 2008 May;43(5):443-50. doi: 10.1002/ppul.20782. PMID 18383112
- [Result] Hamvas A, Heins HB, Guttentag SH, Wegner DJ, Trusgnich MA, Bennet KW, Yang P, Carlson CS, An P, Cole FS. Developmental and genetic regulation of human surfactant protein B in vivo. Neonatology. 2009;95(2):117-24. doi: 10.1159/000153095. Epub 2008 Sep 6. PMID 18776725
- [Result] Druley TE, Vallania FL, Wegner DJ, Varley KE, Knowles OL, Bonds JA, Robison SW, Doniger SW, Hamvas A, Cole FS, Fay JC, Mitra RD. Quantification of rare allelic variants from pooled genomic DNA. Nat Methods. 2009 Apr;6(4):263-5. doi: 10.1038/nmeth.1307. Epub 2009 Mar 1. PMID 19252504
- [Result] Hamvas A, Nogee LM, Wegner DJ, Depass K, Christodoulou J, Bennetts B, McQuade LR, Gray PH, Deterding RR, Carroll TR, Kammesheidt A, Kasch LM, Kulkarni S, Cole FS. Inherited surfactant deficiency caused by uniparental disomy of rare mutations in the surfactant protein-B and ATP binding cassette, subfamily a, member 3 genes. J Pediatr. 2009 Dec;155(6):854-859.e1. doi: 10.1016/j.jpeds.2009.06.006. Epub 2009 Aug 3. PMID 19647838
- [Result] Tomazela DM, Patterson BW, Hanson E, Spence KL, Kanion TB, Salinger DH, Vicini P, Barret H, Heins HB, Cole FS, Hamvas A, MacCoss MJ. Measurement of human surfactant protein-B turnover in vivo from tracheal aspirates using targeted proteomics. Anal Chem. 2010 Mar 15;82(6):2561-7. doi: 10.1021/ac1001433. PMID 20178338
- [Result] Wambach JA, Yang P, Wegner DJ, An P, Hackett BP, Cole FS, Hamvas A. Surfactant protein-C promoter variants associated with neonatal respiratory distress syndrome reduce transcription. Pediatr Res. 2010 Sep;68(3):216-20. doi: 10.1203/PDR.0b013e3181eb5d68. PMID 20539253
- [Result] Anadkat JS, Kuzniewicz MW, Chaudhari BP, Cole FS, Hamvas A. Increased risk for respiratory distress among white, male, late preterm and term infants. J Perinatol. 2012 Oct;32(10):780-5. doi: 10.1038/jp.2011.191. Epub 2012 Jan 5. PMID 22222548
- [Result] Agrawal A, Hamvas A, Cole FS, Wambach JA, Wegner D, Coghill C, Harrison K, Nogee LM. An intronic ABCA3 mutation that is responsible for respiratory disease. Pediatr Res. 2012 Jun;71(6):633-7. doi: 10.1038/pr.2012.21. Epub 2012 Feb 15. PMID 22337229
- [Result] Bereman MS, Tomazela DM, Heins HS, Simonato M, Cogo PE, Hamvas A, Patterson BW, Cole FS, MacCoss MJ. A method to determine the kinetics of multiple proteins in human infants with respiratory distress syndrome. Anal Bioanal Chem. 2012 Jun;403(8):2397-402. doi: 10.1007/s00216-012-5953-3. Epub 2012 Apr 14. PMID 22526637
- [Result] Wambach JA, Wegner DJ, Depass K, Heins H, Druley TE, Mitra RD, An P, Zhang Q, Nogee LM, Cole FS, Hamvas A. Single ABCA3 mutations increase risk for neonatal respiratory distress syndrome. Pediatrics. 2012 Dec;130(6):e1575-82. doi: 10.1542/peds.2012-0918. Epub 2012 Nov 19. PMID 23166334
- [Result] Hamvas A, Deterding RR, Wert SE, White FV, Dishop MK, Alfano DN, Halbower AC, Planer B, Stephan MJ, Uchida DA, Williames LD, Rosenfeld JA, Lebel RR, Young LR, Cole FS, Nogee LM. Heterogeneous pulmonary phenotypes associated with mutations in the thyroid transcription factor gene NKX2-1. Chest. 2013 Sep;144(3):794-804. doi: 10.1378/chest.12-2502. PMID 23430038
- [Result] Sen P, Yang Y, Navarro C, Silva I, Szafranski P, Kolodziejska KE, Dharmadhikari AV, Mostafa H, Kozakewich H, Kearney D, Cahill JB, Whitt M, Bilic M, Margraf L, Charles A, Goldblatt J, Gibson K, Lantz PE, Garvin AJ, Petty J, Kiblawi Z, Zuppan C, McConkie-Rosell A, McDonald MT, Peterson-Carmichael SL, Gaede JT, Shivanna B, Schady D, Friedlich PS, Hays SR, Palafoll IV, Siebers-Renelt U, Bohring A, Finn LS, Siebert JR, Galambos C, Nguyen L, Riley M, Chassaing N, Vigouroux A, Rocha G, Fernandes S, Brumbaugh J, Roberts K, Ho-Ming L, Lo IF, Lam S, Gerychova R, Jezova M, Valaskova I, Fellmann F, Afshar K, Giannoni E, Muhlethaler V, Liang J, Beckmann JS, Lioy J, Deshmukh H, Srinivasan L, Swarr DT, Sloman M, Shaw-Smith C, van Loon RL, Hagman C, Sznajer Y, Barrea C, Galant C, Detaille T, Wambach JA, Cole FS, Hamvas A, Prince LS, Diderich KE, Brooks AS, Verdijk RM, Ravindranathan H, Sugo E, Mowat D, Baker ML, Langston C, Welty S, Stankiewicz P. Novel FOXF1 mutations in sporadic and familial cases of alveolar capillary dysplasia with misaligned pulmonary veins imply a role for its DNA binding domain. Hum Mutat. 2013 Jun;34(6):801-11. doi: 10.1002/humu.22313. Epub 2013 Apr 12. PMID 23505205
- [Result] Wambach JA, Casey AM, Fishman MP, Wegner DJ, Wert SE, Cole FS, Hamvas A, Nogee LM. Genotype-phenotype correlations for infants and children with ABCA3 deficiency. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1538-43. doi: 10.1164/rccm.201402-0342OC. PMID 24871971
- [Result] Wambach JA, Wegner DJ, Heins HB, Druley TE, Mitra RD, Hamvas A, Cole FS. Synonymous ABCA3 variants do not increase risk for neonatal respiratory distress syndrome. J Pediatr. 2014 Jun;164(6):1316-21.e3. doi: 10.1016/j.jpeds.2014.02.021. Epub 2014 Mar 20. PMID 24657120
- [Result] Jackson T, Wegner DJ, White FV, Hamvas A, Cole FS, Wambach JA. Respiratory failure in a term infant with cis and trans mutations in ABCA3. J Perinatol. 2015 Mar;35(3):231-2. doi: 10.1038/jp.2014.236. PMID 25712598
- [Result] Coghlan MA, Shifren A, Huang HJ, Russell TD, Mitra RD, Zhang Q, Wegner DJ, Cole FS, Hamvas A. Sequencing of idiopathic pulmonary fibrosis-related genes reveals independent single gene associations. BMJ Open Respir Res. 2014 Dec 10;1(1):e000057. doi: 10.1136/bmjresp-2014-000057. eCollection 2014. PMID 25553246
- [Result] Ramos EI, Bien-Willner GA, Li J, Hughes AE, Giacalone J, Chasnoff S, Kulkarni S, Parmacek M, Cole FS, Druley TE. Genetic variation in MKL2 and decreased downstream PCTAIRE1 expression in extreme, fatal primary human microcephaly. Clin Genet. 2014 May;85(5):423-32. doi: 10.1111/cge.12197. Epub 2013 Jun 18. PMID 23692340
- [Result] van Meel E, Wegner DJ, Cliften P, Willing MC, White FV, Kornfeld S, Cole FS. Rare recessive loss-of-function methionyl-tRNA synthetase mutations presenting as a multi-organ phenotype. BMC Med Genet. 2013 Oct 8;14:106. doi: 10.1186/1471-2350-14-106. PMID 24103465
- [Result] Szafranski P, Dharmadhikari AV, Wambach JA, Towe CT, White FV, Grady RM, Eghtesady P, Cole FS, Deutsch G, Sen P, Stankiewicz P. Two deletions overlapping a distant FOXF1 enhancer unravel the role of lncRNA LINC01081 in etiology of alveolar capillary dysplasia with misalignment of pulmonary veins. Am J Med Genet A. 2014 Aug;164A(8):2013-9. doi: 10.1002/ajmg.a.36606. Epub 2014 May 19. PMID 24842713
- [Result] Chen YJ, Wambach JA, DePass K, Wegner DJ, Chen SK, Zhang QY, Heins H, Cole FS, Hamvas A. Population-based frequency of surfactant dysfunction mutations in a native Chinese cohort. World J Pediatr. 2016 May;12(2):190-5. doi: 10.1007/s12519-015-0047-x. Epub 2015 Nov 7. PMID 26547207
- [Result] Shen CL, Zhang Q, Meyer Hudson J, Cole FS, Wambach JA. Genetic Factors Contribute to Risk for Neonatal Respiratory Distress Syndrome among Moderately Preterm, Late Preterm, and Term Infants. J Pediatr. 2016 May;172:69-74.e2. doi: 10.1016/j.jpeds.2016.01.031. Epub 2016 Feb 28. PMID 26935785
- [Result] Wambach JA, Yang P, Wegner DJ, Heins HB, Kaliberova LN, Kaliberov SA, Curiel DT, White FV, Hamvas A, Hackett BP, Cole FS. Functional Characterization of ATP-Binding Cassette Transporter A3 Mutations from Infants with Respiratory Distress Syndrome. Am J Respir Cell Mol Biol. 2016 Nov;55(5):716-721. doi: 10.1165/rcmb.2016-0008OC. PMID 27374344
- [Result] Eldridge WB, Zhang Q, Faro A, Sweet SC, Eghtesady P, Hamvas A, Cole FS, Wambach JA. Outcomes of Lung Transplantation for Infants and Children with Genetic Disorders of Surfactant Metabolism. J Pediatr. 2017 May;184:157-164.e2. doi: 10.1016/j.jpeds.2017.01.017. Epub 2017 Feb 16. PMID 28215425
- [Result] Stout MJ, Demaree D, Merfeld E, Tuuli MG, Wambach JA, Cole FS, Cahill AG. Neonatal Outcomes Differ after Spontaneous and Indicated Preterm Birth. Am J Perinatol. 2018 Apr;35(5):494-502. doi: 10.1055/s-0037-1608804. Epub 2017 Nov 28. PMID 29183099
- [Result] Towe CT, White FV, Grady RM, Sweet SC, Eghtesady P, Wegner DJ, Sen P, Szafranski P, Stankiewicz P, Hamvas A, Cole FS, Wambach JA. Infants with Atypical Presentations of Alveolar Capillary Dysplasia with Misalignment of the Pulmonary Veins Who Underwent Bilateral Lung Transplantation. J Pediatr. 2018 Mar;194:158-164.e1. doi: 10.1016/j.jpeds.2017.10.026. Epub 2017 Dec 1. PMID 29198536
- [Result] Chen YJ, Meyer J, Wambach JA, DePass K, Wegner DJ, Fan X, Zhang QY, Hillary H, Cole FS, Hamvas A. Gene variants of the phosphatidylcholine synthesis pathway do not contribute to RDS in the Chinese population. World J Pediatr. 2018 Feb;14(1):52-56. doi: 10.1007/s12519-017-0109-3. Epub 2018 Feb 6. PMID 29411327
- [Result] Attarian SJ, Leibel SL, Yang P, Alfano DN, Hackett BP, Cole FS, Hamvas A. Mutations in the thyroid transcription factor gene NKX2-1 result in decreased expression of SFTPB and SFTPC. Pediatr Res. 2018 Sep;84(3):419-425. doi: 10.1038/pr.2018.30. Epub 2018 Apr 11. PMID 29538355
- [Result] Thomas BJ, Wight IE, Chou WYY, Moreno M, Dawson Z, Homayouni A, Huang H, Kim H, Jia H, Buland JR, Wambach JA, Cole FS, Pak SC, Silverman GA, Luke CJ. CemOrange2 fusions facilitate multifluorophore subcellular imaging in C. elegans. PLoS One. 2019 Mar 26;14(3):e0214257. doi: 10.1371/journal.pone.0214257. eCollection 2019. PMID 30913273
- [Result] Wambach JA, Yang P, Wegner DJ, Heins HB, Luke C, Li F, White FV, Cole FS. Functional Genomics of ABCA3 Variants. Am J Respir Cell Mol Biol. 2020 Oct;63(4):436-443. doi: 10.1165/rcmb.2020-0034MA. PMID 32692933
- [Result] Alysandratos KD, Russo SJ, Petcherski A, Taddeo EP, Acin-Perez R, Villacorta-Martin C, Jean JC, Mulugeta S, Rodriguez LR, Blum BC, Hekman RM, Hix OT, Minakin K, Vedaie M, Kook S, Tilston-Lunel AM, Varelas X, Wambach JA, Cole FS, Hamvas A, Young LR, Liesa M, Emili A, Guttentag SH, Shirihai OS, Beers MF, Kotton DN. Patient-specific iPSCs carrying an SFTPC mutation reveal the intrinsic alveolar epithelial dysfunction at the inception of interstitial lung disease. Cell Rep. 2021 Aug 31;36(9):109636. doi: 10.1016/j.celrep.2021.109636. PMID 34469722